CLINICAL TRIAL: NCT05283720
Title: Phase 1b/2, Open-Label Study to Evaluate Safety and Tolerability of Epcoritamab in Combination With Anti-Neoplastic Agents in Subjects With Non-Hodgkin Lymphoma
Brief Title: A Study to Evaluate Adverse Events and Change in Disease Activity of Subcutaneous (SC) Epcoritamab in Combination With Oral and Intravenous Anti-Neoplastic Agents in Adult Participants With Non-Hodgkin Lymphoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Genmab (Industry)
Collaborators: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: M22-132; 2023-505347-38 (Other: EU CT)
Record Dates: First submitted 2022-03-09; First posted 2022-03-17 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Non-Hodgkin Lymphoma
Keywords: Non-Hodgkin Lymphoma; Epcoritamab; Lenalidomide; Ibrutinib; Polatuzumab Vedotin; Rituximab; Cyclophosphamide; Doxorubicin Hydrochloride (HCl]; Prednisone (pola-R-CHP); ABBV-GMAB-3013; Cancer; Relapsed/Refractory (R/R) Diffuse Large B-Cell Lymphoma (DLBCL), Venetoclax,; Venclexta; ABT-199; GDC-0199; CC-99282; EPCORE; Pirtobrutinib; Mantle Cell Lymhoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Leukemia, Hairy Cell; Neoplasms; Recurrence; Lymphoma, Large B-Cell, Diffuse | interventions — Lenalidomide; ibrutinib; Rituximab; Cyclophosphamide; Doxorubicin; Prednisone; polatuzumab vedotin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (13):
- Arm 1: Dose Escalation (Experimental): Participants with relapsed/refractory (R/R) diffuse large B-cell lymphoma (DLBCL) will receive escalating doses of epcoritamab in combination with lenalidomide in 28 day cycles.
  Interventions: Drug: Epcoritamab; Drug: Lenalidomide
- Arm 2: Dose Escalation (Experimental): Participants with R/R DLBCL will receive escalating doses of epcoritamab in combination with ibrutinib and lenalidomide in 28 day cycles.
  Interventions: Drug: Epcoritamab; Drug: Lenalidomide; Drug: Ibrutinib
- Arm 3: Dose Escalation (Experimental): Participants with newly diagnosed treatment-naïve DLBCL will receive escalating doses of epcoritamab in combination with polatuzumab vedotin, rituximab, cyclophosphamide, doxorubicin hydrochloride (HCl), and prednisone (pola-R-CHP) in 21 day cycles.
  Interventions: Drug: Epcoritamab; Drug: Rituximab; Drug: Cyclophosphamide; Drug: Doxorubicin Hydrochloride [HCl]; Drug: Prednisone; Drug: Polatuzumab Vedotin
- Arm 4: Dose Escalation (Experimental): Participants with R/R DLBCL will receive escalating doses of epcoritamab in combination with CC-99282 in 28 day cycles.
  Interventions: Drug: Epcoritamab; Drug: CC-99282
- Arm 5: Dose Escalation (Experimental): Participants with R/R follicular lymphoma (FL) will receive escalating doses of epcoritamab in combination with CC-99282 in 28 day cycles.
  Interventions: Drug: Epcoritamab; Drug: CC-99282
- Arm 6A: Dose Escalation (Experimental): Participants with R/R mantle cell lymphoma (MCL) will receive escalating doses of epcoritamab in combination with ibrutinib in 28 day cycles.
  Interventions: Drug: Epcoritamab; Drug: Ibrutinib
- Arm 1: Dose Expansion (Experimental): Participants with R/R DLBCL will receive the recommended dose of epcoritamab in combination with lenalidomide in 28 day cycles.
  Interventions: Drug: Epcoritamab; Drug: Lenalidomide
- Arm 2: Dose Expansion (Experimental): Participants with R/R DLBCL will receive the recommended dose of epcoritamab in combination with oral ibrutinib and oral lenalidomide in 28 day cycles.
  Interventions: Drug: Epcoritamab; Drug: Lenalidomide; Drug: Ibrutinib
- Arm 3: Dose Expansion (Experimental): Participants newly diagnosed treatment-naïve DLBCL will receive the recommended dose of epcoritamab in combination with polatuzumab vedotin, rituximab, cyclophosphamide, doxorubicin hydrochloride (HCl), and prednisone (pola-R-CHP) in 21 day cycles.
  Interventions: Drug: Epcoritamab; Drug: Rituximab; Drug: Cyclophosphamide; Drug: Doxorubicin Hydrochloride [HCl]; Drug: Prednisone; Drug: Polatuzumab Vedotin
- Arm 3B: Dose Expansion (Experimental): Participants newly diagnosed treatment-naïve DLBCL will receive the recommended dose of epcoritamab in combination with polatuzumab vedotin, rituximab, cyclophosphamide, doxorubicin hydrochloride (HCl), and prednisone (pola-R-CHP), in 21 day cycles,until unacceptable toxicity, withdrawal of consent, or completion of treatment.
  Interventions: Drug: Epcoritamab; Drug: Rituximab; Drug: Cyclophosphamide; Drug: Doxorubicin Hydrochloride [HCl]; Drug: Prednisone; Drug: Polatuzumab Vedotin
- Arm 4: Dose Expansion (Experimental): Participants with R/R DLBCL will receive the recommended dose of epcoritamab in combination with CC-99282 in 28 day cycles.
  Interventions: Drug: Epcoritamab; Drug: CC-99282
- Arm 5: Dose Expansion (Experimental): Participants with R/R FL will receive the recommended dose of epcoritamab in combination with CC-99282 in 28 day cycles.
  Interventions: Drug: Epcoritamab; Drug: CC-99282
- Arm 6: Dose Expansion (Experimental): Participants with R/R MCL will receive the recommended dose of epcoritamab in combination with ibrutinib in 28 day cycles.
  Interventions: Drug: Epcoritamab; Drug: Ibrutinib

INTERVENTIONS:
Drug: Epcoritamab — Subcutaneous Injection (SC)
  Other Names: ABBV-GMAB-3013;
Drug: Lenalidomide — Oral; Capsule
  Arms: Arm 1: Dose Escalation; Arm 1: Dose Expansion; Arm 2: Dose Escalation; Arm 2: Dose Expansion
Drug: Ibrutinib — Oral; Capsule
  Other Names: Imbruvica
  Arms: Arm 2: Dose Escalation; Arm 2: Dose Expansion; Arm 6: Dose Expansion; Arm 6A: Dose Escalation
Drug: Rituximab — Intravenous (IV); Injection
  Arms: Arm 3: Dose Escalation; Arm 3: Dose Expansion; Arm 3B: Dose Expansion
Drug: Cyclophosphamide — IV; Injection
  Arms: Arm 3: Dose Escalation; Arm 3: Dose Expansion; Arm 3B: Dose Expansion
Drug: Doxorubicin Hydrochloride [HCl] — IV; Injection
  Arms: Arm 3: Dose Escalation; Arm 3: Dose Expansion; Arm 3B: Dose Expansion
Drug: Prednisone — Oral; Tablet
  Arms: Arm 3: Dose Escalation; Arm 3: Dose Expansion; Arm 3B: Dose Expansion
Drug: Polatuzumab Vedotin — IV; Injection
  Arms: Arm 3: Dose Escalation; Arm 3: Dose Expansion; Arm 3B: Dose Expansion
Drug: CC-99282 — Oral; Capsule
  Arms: Arm 4: Dose Escalation; Arm 4: Dose Expansion; Arm 5: Dose Escalation; Arm 5: Dose Expansion

SUMMARY:
B-cell Lymphoma is an aggressive and rare cancer of a type of immune cell (a white blood cell responsible for fighting infections). The purpose of this study is to assess the safety and tolerability of epcoritamab in combination with anti-neoplastic agents in adult participants with Non-Hodgkin lymphoma (NHL). Adverse events and change in disease activity will be assessed.

Epcoritamab is an investigational drug being developed for the treatment of NHL. Study doctors put the participants in groups called treatment arms. The combination of epcoritamab with anti-neoplastic agents will be explored. Each treatment arm receives a different treatment combination depending on eligibility. Approximately 496 adult participants with NHL will be enrolled in 100 sites globally.

In both the dose escalation and dose expansion arms participants will receive subcutaneous (SC) epcoritamab in 28 day, 21 day, or 56 day cycles dependent on the arm in combination with the anti-neoplastic agents described below:

1: Oral lenalidomide in participants (PPTS) with relapsed/refractory (R/R) diffuse large B-cell lymphoma (DLBCL); 2: Oral ibrutinib and oral lenalidomide in PPTS with R/R DLBCL; 3: Intravenous (IV) polatuzumab vedotin, IV rituximab, IV cyclophosphamide, IV doxorubicin hydrochloride (HCl), and oral prednisone (pola-R-CHP) in PPTS with newly diagnosed treatment-naïve DLBCL, or completion of treatment in 3B; 4: Oral CC-99282 in PPTS with R/R DLBCL; 5: Oral CC-99282 in PPTS with R/R follicular lymphoma (FL); 6A: Oral ibrutinib in PPTS with R/R mantle cell lymphoma (MCL).

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the study at an approved institution (hospital or clinic). The effect of the treatment will be frequently checked by medical assessments, blood tests, questionnaires and side effects.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of:

  -- Diffuse large B-cell lymphoma (DLBCL) (de novo or histologically transformed from follicular lymphoma (FL) or nodal marginal zone lymphoma) with histologically confirmed CD20+ disease, inclusive of the following according to World Health Organization (WHO) 2016 classification and documented in pathology report:
  * DLBCL, not otherwise specified (NOS).
  * High-grade B cell lymphoma with MYC and BCL-2 and/or BCL-6 translocations per WHO 2016 ("double-hit" or "triple-hit") Note: High-grade B-cell lymphomas NOS or other double- /triple-hit lymphomas (with histologies not consistent with DLBCL) are not eligible.
  * Follicular lymphoma (FL) Grade 3B. OR
* FL with histologically confirmed CD20+ Grade 1 to 3a and no evidence of histologic transformation to an aggressive lymphoma at most recent representative tumor biopsy, according to WHO 2016 classification. OR
* Mantle cell lymphoma (MCL) with histologically confirmed CD20+ disease at most recent representative tumor biopsy according to the WHO 2016 classification with evidence of overexpression of cyclin D1 in association with relevant markers or evidence of t(11;14) assessed by flow cytometry, fluorescence in situ hybridization (FISH), or polymerase chain reaction (PCR).
* Eastern Cooperative Oncology Group (ECOG) performance status 0 - 2, except for Arm 6A where ECOG performance status must be 0-1.
* Must have 1 or more measurable disease sites:

  * A positron emission tomography (PET) /computed tomography (CT) scan demonstrating PET-positive lesion(s) AND
  * At least 1 measurable nodal lesion (long axis > 1.5 cm) or >= 1 measurable extra-nodal lesion (long axis > 1.0 cm) on CT scan or magnetic resonance imaging (MRI).

Exclusion Criteria:

* Prior treatment with epcoritamab or any other bispecific antibody targeting CD3 and CD20.
* Toxicities from prior anticancer therapy that have not resolved to Common Terminology Criteria for Adverse Events (CTCAE, v 5.0), Grade 2 or below, with the exception of alopecia. Other eligibility criteria (e.g., laboratory, cardiac criteria) must also be met.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 496 (Estimated)
Dates: Start 2022-06-14 (Actual); Primary Completion 2032-11 (Estimated); Study Completion 2032-11 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Dose-Limiting Toxicities (DLT) | Up to Approximately 5 Years
  DLT events are defined as clinically significant adverse events or abnormal laboratory values assessed as unrelated to disease progression, underlying disease, intercurrent illness, or concomitant medications.

SECONDARY OUTCOMES:
Best Overall Response (BOR) per Investigator | Up to Approximately 5 Years
  BOR is defined as the percentage of participants who achieved best overall response of CR or PR by Lugano 2014 criteria as assessed by the investigator.
Duration of response (DOR) per Investigator | Up to Approximately 5 Years
  DOR is defined for participants who achieved best overall response of CR or PR ('responders'), as the time in months from initial CR/PR to the earliest occurrence of radiographic progression determined by Lugano 2014 criteria as assessed by the investigator, or death from any cause.
Number of Participants with Progression-free survival (PFS) | Up to Approximately 5 Years
  PFS is defined as the time in months from the first dose of study drug to the earliest occurrence of disease progression determined by Lugano 2014 criteria as assessed by investigator, or death from any cause.
Percentage of Participants with Complete Response (CR) | Up to Approximately 5 Years
  CR is defined as the percentage of participantswho achieved best overall response of CR determined by Lugano 2014 criteria as assessed by investigator.
Time-to-response (TTR) | Up to Approximately 5 Years
  TTR is defined as the number of months from the date of first dose to the date of best overall response of CR or PR ('responders') determined by Lugano 2014 criteria as assessed by investigator.
Time to Next Antilymphoma Therapy (TTNT) | Up to Approximately 5 Years
  Time to next antilymphoma therapy.
Rate of Minimal Residual Disease (MRD) Negativity | Up to Approximately 5 Years
  MRD is defined as the percentage of participants with assessment of the minimal residual disease.
Overall Survival (OS) | Up to Approximately 5 Years
  (OS) is defined as the time in months from first dose of epcoritamab to death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (75):
- United States (18):
  - The University of Arizona Cancer Center - North Campus /ID# 242219, Tucson, Arizona
  - Yale University School of Medicine /ID# 242089, New Haven, Connecticut
  - Christiana Care Health Service /ID# 242301, Newark, Delaware
  - Tampa General Hospital /ID# 246748, Tampa, Florida
  - Winship Cancer Institute of Emory University /ID# 242153, Atlanta, Georgia
  - University of Maryland, Baltimore /ID# 242218, Baltimore, Maryland
  - Alliance for Multispecialty Research (AMR) - Kansas City /ID# 242144, Kansas City, Missouri
  - Northwell Health - Monter Cancer Center /ID# 245435, Lake Success, New York
  - Icahn School of Medicine at Mount Sinai /ID# 242123, New York, New York
  - Novant Health Presbyterian Medical Center /ID# 242148, Charlotte, North Carolina
  - East Carolina University - Brody School of Medicine /ID# 242506, Greenville, North Carolina
  - Novant Health Forsyth Medical Center /ID# 242198, Winston-Salem, North Carolina
  - Thomas Jefferson University Hospital /ID# 242077, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center /ID# 242106, Philadelphia, Pennsylvania
  - Thompson Cancer Survival Ctr /ID# 242150, Knoxville, Tennessee
  - Joe Arrington Cancer Research /ID# 242226, Lubbock, Texas
  - Swedish Cancer Institute /ID# 242269, Seattle, Washington
  - MultiCare Institute for Research & Innovation /ID# 242127, Tacoma, Washington
- Beijing Cancer Hospital /ID# 252303, Beijing, Beijing Municipality, China
- Czechia (4):
  - Fakultní Nemocnice Brno - Jihlavská /ID# 242683, Brno, Brno-mesto
  - Fakultní nemocnice Hradec Králové - Sokolská /ID# 241722, Hradec Králové, Hradec Kralove
  - Fakultni Nemocnice Ostrava /ID# 242684, Ostrava, Ostrava-mesto
  - Vseobecna Fakultni Nemocnice v Praze /ID# 242685, Prague, Praha 17
- Denmark (2):
  - Aarhus Universitetshospital - Skejby /ID# 242670, Aarhus, Central Jutland
  - Aalborg University Hospital /ID# 242734, Aalborg, North Denmark
- France (10):
  - CHU Clermont-Ferrand /ID# 242344, Clermont, Auvergne-Rhône-Alpes
  - CHU de Rennes - PONTCHAILLOU /ID# 242339, Rennes, Brittany Region
  - Centre Hospitalier Régional Universitaire de Nancy - Hôpitaux de Brabois /ID# 242342, Vandœuvre-lès-Nancy, Meurthe-et-Moselle
  - CHRU Lille - Hopital Claude Huriez /ID# 242335, Lille, Nord
  - IUCT Oncopole /ID# 242340, Toulouse, Occitanie
  - Hopitaux Universitaires Henri Mondor - Hopital Henri Mondor /ID# 242337, Créteil, Paris
  - Centre Hospitalier Universitaire de Nantes, Hotel Dieu -HME /ID# 242345, Nantes, Pays de la Loire Region
  - HCL - Hopital Lyon Sud /ID# 242349, Pierre-Bénite, Rhone
  - Hôpital Saint-Louis /ID# 242336, Paris
  - Hopital Pitie Salpetriere /ID# 242343, Paris, Île-de-France Region
- Germany (6):
  - Universitaetsklinikum Ulm /ID# 244265, Ulm, Baden-Wurttemberg
  - Klinikum Augsburg /ID# 244523, Augsburg, Bavaria
  - Universitaetsklinikum Wuerzburg /ID# 245453, Würzburg, Bavaria
  - Universitaetsklinikum Giessen und Marburg /ID# 245308, Marburg, Hesse
  - Universitaetsklinikum Leipzig /ID# 245513, Leipzig, Saxony
  - Universitaetsklinikum Regensburg /ID# 244517, Regensburg
- Hungary (4):
  - Debreceni Egyetem-Klinikai Kozpont /ID# 242450, Debrecen, Hajdú-Bihar
  - Somogy Varmegyei Kaposi Mor Oktato Korhaz /ID# 245935, Kaposvár, Somogy County
  - Semmelweis Egyetem /ID# 242454, Budapest
  - Orszagos Onkologiai Intezet /ID# 242458, Budapest
- Israel (4):
  - Hadassah Medical Center-Hebrew University /ID# 243013, Jerusalem, Jerusalem
  - The Chaim Sheba Medical Center /ID# 243010, Ramat Gan, Tel Aviv
  - Tel Aviv Sourasky Medical Center /ID# 243012, Tel Aviv, Tel Aviv
  - Rabin Medical Center. /ID# 243014, Petah Tikva
- Japan (3):
  - Hokkaido University Hospital /ID# 248999, Sapporo, Hokkaido
  - Kyoto University Hospital /ID# 248997, Kyoto, Kyoto
  - National Cancer Center Hospital /ID# 248995, Chuo-ku, Tokyo
- Netherlands (5):
  - Maastricht Universitair Medisch Centrum /ID# 243317, Maastricht, Limburg
  - Vrije Universiteit Medisch Centrum /ID# 243319, Amsterdam, North Holland
  - Leids Universitair Medisch Centrum /ID# 243316, Leiden, South Holland
  - Duplicate_Erasmus Medisch Centrum /ID# 243315, Rotterdam, South Holland
  - Universitair Medisch Centrum Groningen /ID# 243318, Groningen
- South Korea (5):
  - Seoul National University Bundang Hospital /ID# 242404, Seongnam-si, Gyeonggido
  - Seoul National University Hospital /ID# 242402, Seoul, Seoul Teugbyeolsi
  - Asan Medical Center /ID# 242400, Seoul, Seoul Teugbyeolsi
  - Samsung Medical Center /ID# 242401, Seoul, Seoul Teugbyeolsi
  - The Catholic University of Korea, Seoul St. Marys Hospital /ID# 242403, Seoul, Seoul Teugbyeolsi
- Spain (10):
  - Instituto Catalan de Oncologia (ICO) Badalona /ID# 243265, Badalona, Barcelona
  - Institut Català d'Oncologia (ICO) - L'Hospitalet /ID# 243261, L'Hospitalet de Llobregat, Barcelona
  - Clinica Universidad de Navarra - Pamplona /ID# 245031, Pamplona, Navarre
  - Hospital Universitario Vall de Hebron /ID# 243260, Barcelona
  - CLINICA UNIVERSIDAD DE NAVARRA-Madrid /ID# 243268, Madrid
  - Hospital Universitario Fundacion Jimenez Diaz /ID# 243264, Madrid
  - Hospital Universitario 12 de Octubre /ID# 243262, Madrid
  - Hospital Universitario de Salamanca /ID# 243368, Salamanca
  - Hospital Universitario Virgen del Rocio /ID# 243267, Seville
  - Hospital Clinico Universitario de Valencia /ID# 243269, Valencia
- Taiwan (3):
  - China Medical University Hospital /ID# 242893, Taichung
  - National Cheng Kung University Hospital /ID# 242894, Tainan
  - Taipei Veterans General Hosp /ID# 242892, Taipei

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols, analyses plans, clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M22-132